CLINICAL TRIAL: NCT03877029
Title: Long-term Effects Following Treatment of Women With Screen-detected Versus Symptomatic Breast Cancer
Brief Title: Long-term Effects of Breast Cancer Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: The Dam Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/FO244363
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Mammography; Breast cancer screening; Health related quality of life; Long-term effects of breast cancer treatment; Screen-detected breast cancer; Symptomatic breast cancer; Tumor characteristics; Interval breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study II: * Women with a screen-detected breast cancer after attending BreastScreen Norway
  * Women with symptomatic breast cancer, who have never been screened in BreastScreen Norway
  * Women with interval breast cancer after attending BreastScreen Norway
  * Women free from breast cancer
- Study III: * Women with a screen-detected breast cancer after attending BreastScreen Norway
  * Women with interval breast cancer after attending BreastScreen Norway and women with symptomatic breast cancer, who have never been screened in BreastScreen Norway

SUMMARY:
The objective of this project is to generate evidence about quality of life related to side effects of treatment of women with screen-detected versus symptomatic breast cancer. The project will investigate the impact of detection mode (by screening or by symptoms) versus tumor characteristics as a predictor of quality of life among breast cancer survivors. The burden of long-term effects, measured as quality of life at specific points after diagnosis, will be compared between these groups. The results will also be compared with a control group of women, who have attended screening, but never been diagnosed with breast cancer.

DETAILED DESCRIPTION:
The project will include a retrospective information which will be collected by using a self-administered questionnaire about the treatment women received and their quality of life at certain time points after a breast cancer diagnosis. Women aged 50-69 years at the time of diagnosis are the target group of BreastScreen Norway and also for this project.

The women will be identified from the Cancer Registry databases. The questionnaire will be based on EQ-5D-5L and will be developed in close collaboration with breast cancer survivors who have personally experienced the long-term effects of breast cancer treatment, whether resulting from screen-detected or symptomatic breast cancer.

The questionnaire will cover topics related to demographics, treatment, and information required to estimate health related quality of life (HRQoL) and quality-adjusted life years (QALY). Information about detection mode and disease stage at diagnosis will be extracted from the Cancer Registry.

Study I - a review of the literature in a paper describing and analyzing the current evidence on quality of life among women diagnosed with breast cancer and treated for this disease, with a focus on disease stage at diagnosis. Due to substantial changes in treatment during the last decades, only studies reporting on women who have received treatment in 1995 or later will be included. Solely studies written in English will be included.

For studies II and III, data collected from the self-administered questionnaire will be used. In addition, information about screening history and tumor characteristics will be obtained from the Cancer Registry of Norway.

In Study II, quality of life will be compared between about 1000 women treated for screen-detected, about 1000 women treated for symptomatic, about 1000 women treated for interval cancer and about 1000 women without any diagnosis of breast cancer. The main hypothesis is that women with screen-detected breast cancer have a higher quality of life than women diagnosed with symptomatic breast cancer.

Study III will be a continuation of Study II, and will aim to investigate the impact of detection mode versus tumor characteristics and treatment types as the main predictor of long-term quality of life among women diagnosed and treated for breast cancer among the two groups of women, those diagnosed with screen-detected breast cancer versus those diagnosed with interval breast and symptomatic breast cancer.

ELIGIBILITY:
Study II

Inclusion Criteria:

* Screened in BreastScreen Norway and diagnosed with breast cancer between 2006 and 2017
* Diagnosed with symptomatic breast cancer between 2006 and 2017 and never attended screening
* Screened in BreastScreen Norway and diagnosed with interval breast cancer between 2006 and 2017
* Screened in BreastScreen Norway and have never been diagnosed with breast cancer

Exclusion Criteria:

* Death after recruitment

Study III

Inclusion Criteria:

* Screened in BreastScreen Norway and diagnosed with breast cancer between 2006 and 2017
* Screened in BreastScreen Norway and diagnosed with interval breast cancer between 2006 and 2017
* Diagnosed with symptomatic breast cancer between 2006 and 2017 and never attended screening

Exclusion Criteria:

* Death after recruitment

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include women residing in Norway, who are currently alive and were invited and attended, and were invited but did not attend the screening program. Among the attending and not attending women, women who were diagnosed with breast cancer 2006-2017 will be randomly selected. The women diagnosed with breast cancer will be stratified by detection mode (screen-detected versus symptomatic breast cancer). The women within each group will be matched by age. Additionally, women who have never had a diagnosis of breast cancer will be randomly selected from the target population of BreastScreen Norway.
Sampling Method: Non-Probability Sample
Enrollment: 4487 (Actual)
Dates: Start 2019-11-23 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Quality of life score | 2006-2017
  Quality of life measure from 0 to 100 on a visual analogue scale
QALY (Quality-Adjusted-Life-Year) | 2006-2017
  QALY is calculated by estimating the years of life remaining for a woman following a particular treatment or intervention and weighting each year with her corresponding health related quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Hofvind, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Cancer Registry of Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moshina N, Falk RS, Hofvind S. Long-term quality of life among breast cancer survivors eligible for screening at diagnosis: a systematic review and meta-analysis. Public Health. 2021 Oct;199:65-76. doi: 10.1016/j.puhe.2021.08.008. Epub 2021 Sep 21. PMID 34560477